CLINICAL TRIAL: NCT05683873
Title: Stroke-induced Myocardial Dysfunction: Role of GDF-15 (SMOG-15) Clinical Work Package
Acronym: SMOG-15
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BEJOT ANR 2019
Record Dates: First submitted 2023-01-02; First posted 2023-01-13 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Osteoprotegerin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Electrocardiogram — Inclusion visit, V1, V2 and V3
Procedure: transthoracic echocardiography — V1, V2 and V3
Biological: standard biology — Inclusion visit
Biological: determination of serum GDF-15, osteoprotegerin and ST-2 — Inclusion visit, V1, V2 and V3
Biological: Ultrasensitive Troponin-Ic — Inclusion visit, V1, V2 and V3
Other: Collection of clinical and radiological data — Inclusion visit, V1 and V3: clinical data only V2: clinical and radiological data
Other: 72-hour continuous Holter-ECG recording — V1

SUMMARY:
The aim of this study is to analyze the relationship between the blood biomarker GDF-15 and heart damage after stroke.

It is being conducted in France, in the Neurology Department of the Dijon University Hospital (Burgundy). The research is interventional because a biological blood test will be performed, as well as a heart rhythm recording and several cardiac echograms during the hospitalization of the participants and during the follow-up consultation scheduled 4 to 6 months after the stroke.

A total of 130 stroke patients will participate in this study.

Participation includes 4 visits:

* Inclusion visit (within 24 hours of the first stroke symptoms)
* visit 1 (within 24 to 72 hours of stroke)
* visit 2 (within 48 hours of visit 1)
* Visit 3 (approximately 4-6 months post-stroke)

ELIGIBILITY:
Inclusion Criteria:

* Adult with acute symptomatic cerebral infarction documented by brain imaging on admission (cerebral angioscan or cerebral MRI)
* Whose first symptoms appeared within 24 hours before inclusion
* Whose consent to participate in this study was obtained from the patient or a close relative.

Exclusion Criteria:

* Person with a history of symptomatic stroke, either ischemic or hemorrhagic
* Anyone with a history of heart disease including: atrial fibrillation or flutter (known or discovered on admission), chronic heart failure, pacemaker, defibrillator, or other cardiac devices
* Person with acute heart failure, suspected infective endocarditis, STEMI, or concurrent pulmonary embolism
* A person who is not a member or beneficiary of a social security system
* Person deprived of liberty
* Person subject to a legal protection measure (curatorship, guardianship)
* Person subject to a legal protection measure
* Pregnant, parturient or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-02-13 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Global Longitudinal Strain (GLS) of the left ventricle measured by trans-thoracic ultrasound (TTE) | within 24 to 72 hours post-stroke

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

IPD SHARING:
Plan to Share IPD: No